CLINICAL TRIAL: NCT07167368
Title: Efficacy and Safety of Home-Based Exercise Rehabilitation in Patients With Cardiorenal Syndrome Complicated by Chronic Heart Failure With Reduced Ejection Fraction (HFrEF): A Randomized Controlled Trial
Brief Title: Exercise Rehabilitation for Cardiorenal Syndrome in HFrEF Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haiyan Pan (Other)
Responsible Party: Sponsor-Investigator, Haiyan Pan, Professor and Chief Physician, Department of Cardiology, Affiliated Hospital of Nantong University
Organization: Affiliated Hospital of Nantong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-K124-01-B
Record Dates: First submitted 2025-08-18; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Cardiorenal Syndrome
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic Treatment Group (Active Comparator): Patients with HFrEF and chronic kidney dysfunction receive 6 months of basic drug treatment, with regular follow-up during the period.
  Interventions: Drug: Standardized Basic Drug Therapy for HFrEF with Chronic Kidney Dysfunction
- Exercise Rehabilitation Group (Experimental): Patients with HFrEF and chronic kidney dysfunction receive 6 months of basic drug treatment combined with home-based exercise rehabilitation. Exercise prescriptions are formulated based on cardiopulmonary exercise test results (using heart rate at anaerobic threshold) or 6MWT (for those unable to complete cardiopulmonary exercise tests), with follow-up conducted throughout the period.
  Interventions: Drug: Standardized Basic Drug Therapy for HFrEF with Chronic Kidney Dysfunction; Behavioral: Home-based Personalized Exercise Rehabilitation

INTERVENTIONS:
Drug: Standardized Basic Drug Therapy for HFrEF with Chronic Kidney Dysfunction — Participants receive standardized basic drug therapy for HFrEF and chronic kidney dysfunction in accordance with clinical practice guidelines. Medications include but are not limited to angiotensin-converting enzyme inhibitors (ACEIs), angiotensin receptor blockers (ARBs), beta-blockers, mineralocorticoid receptor antagonists (MRAs), and diuretics, with dosage adjustments based on individual patient conditions.
  Other Names: Guideline-Based Basic Medication Regimen for CRS Patients with HFrEF
Behavioral: Home-based Personalized Exercise Rehabilitation — On the basis of basic drug treatment, participants in the exercise rehabilitation group receive personalized home-based exercise prescriptions. Prescriptions are developed according to cardiopulmonary exercise test results (using heart rate at anaerobic threshold) or 6MWT (for those unable to complete cardiopulmonary exercise tests). The 6-month exercise program includes aerobic exercises (e.g., brisk walking, cycling), with intensity, duration, and frequency adjusted based on individual tolerance and progress.
  Other Names: Home-Centered Customized Exercise Program for CRS with HFrEF
  Arms: Exercise Rehabilitation Group

SUMMARY:
This study aims to investigate the efficacy and safety of exercise rehabilitation in patients with cardiorenal syndrome (CRS).

Building on previous research demonstrating that exercise rehabilitation can effectively improve cardiac function and cardiopulmonary endurance in patients with chronic heart failure, this study will further explore its role in the context of CRS, a condition where such effects remain understudied. CRS patients typically exhibit reduced cardiopulmonary endurance, with significantly lower peak oxygen uptake (VO₂ peak) and 6-minute walk test (6MWT) distance compared to non-CRS patients.

Adults aged 18-75 with chronic heart failure with reduced ejection fraction (HFrEF) complicated by chronic renal insufficiency will be enrolled and randomly assigned to two groups: 1. Basic treatment group: 30 patients receive only basic drug treatment for 6 months. 2. Exercise rehabilitation group: 30 patients receive basic drug treatment combined with home-based exercise rehabilitation for 6 months (with personalized exercise prescriptions formulated based on cardiopulmonary exercise test results or 6MWT for those unable to complete the former). The study will explore the efficacy and safety of exercise rehabilitation in the prevention and management of CRS by comparing changes in target biomarkers, renal function indicators, cardiac function indicators, cardiopulmonary exercise test results, Minnesota Living with Heart Failure Questionnaire scores, and the incidence of adverse events before and after treatment between the two groups.

The participants will:

Complete cardiopulmonary exercise tests or 6MWT before treatment initiation. Receive basic drug treatment; those in the exercise rehabilitation group will additionally perform home-based exercise rehabilitation according to the exercise prescription.

Attend regular follow-up visits within 6 months. Undergo assessments of related indicators (biomarkers, renal function, cardiac function, etc.) before and after treatment.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of home-based exercise rehabilitation as an adjuvant intervention for patients with Cardiorenal Syndrome (CRS) complicated by Chronic Heart Failure with Reduced Ejection Fraction (HFrEF). Building on prior evidence that exercise rehabilitation improves cardiac function and cardiopulmonary endurance in patients with uncomplicated chronic heart failure, this study addresses a critical gap: the lack of data on how such interventions perform in CRS, a condition characterized by bidirectional cardiorenal impairment that often exacerbates both cardiac and renal dysfunction.

CRS patients with HFrEF typically exhibit reduced cardiopulmonary reserve, as evidenced by lower peak oxygen uptake (VO₂ peak) and 6-minute walk test (6MWT) distance compared to non-CRS patients. This impairment is driven by intertwined pathophysiological mechanisms, including neurohormonal activation, systemic inflammation, and reduced renal clearance of cardiotoxic metabolites-factors that may be modulated by structured exercise. The home-based exercise approach is selected for its clinical relevance: it aligns with long-term patient adherence (avoiding barriers to clinic-based training, such as transportation or scheduling) and allows for personalized intensity adjustments, a key safety consideration in patients with dual organ dysfunction.

Exercise prescriptions for the intervention group are tailored using a two-step assessment protocol to ensure safety and individualization:

1. Cardiopulmonary Exercise Test (CPET): For patients able to complete CPET (per exercise risk assessment), the anaerobic threshold (AT) is identified via gas exchange analysis (using a metabolic cart). Exercise intensity is set at 60-70% of the heart rate corresponding to AT (HR-AT)-a range validated to improve cardiopulmonary endurance without inducing excessive cardiac or renal stress in HFrEF patients.
2. 6MWT Alternative: For patients unable to complete CPET (e.g., due to severe dyspnea or fatigue), exercise intensity is derived from 6MWT results. The target walking speed is set at 70-80% of the average speed achieved during the 6MWT, with duration adjusted to match energy expenditure levels equivalent to the CPET-derived protocol.

The 6-month exercise program focuses on aerobic training (e.g., brisk walking, stationary cycling) with progressive adjustments: initial sessions are 20-30 minutes, 3 times weekly, with 5-10 minute increments in duration (up to 45 minutes) and 5-10% increments in intensity every 2 weeks, based on patient-reported tolerance (assessed via the Borg Rating of Perceived Exertion scale, 0-10) and monthly follow-up monitoring.

To mitigate intervention-related risks, all participants undergo monthly remote or in-clinic follow-up:

* Vital Sign Checks: Resting heart rate, blood pressure, and body weight (to monitor fluid retention, a marker of renal or cardiac decompensation) are recorded at each visit.
* Adverse Event Tracking: Any cardiac (e.g., angina, arrhythmia), renal (e.g., acute kidney injury), or musculoskeletal events are documented using standardized clinical definitions, with protocol adjustments (e.g., temporary exercise pause, intensity reduction) implemented as needed.

This design ensures that the intervention is both mechanistically targeted to CRS pathophysiology and practically feasible for long-term patient engagement, while prioritizing safety in a vulnerable patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronically stable HFrEF complicated by kidney dysfunction (eGFR < 90 mL/min/1.73m²)
* NYHA class II-III
* Low risk in exercise risk assessment
* Aged 18-75 years

Exclusion Criteria:

* Uncontrolled hypertension
* Severe arrhythmias (including frequent ventricular premature contractions, ventricular tachycardia, rapid atrial fibrillation, sick sinus syndrome, and second-degree or higher atrioventricular block)
* Obstructive hypertrophic cardiomyopathy
* Moderate to severe stenotic valvular heart disease
* Deep vein thrombosis or pulmonary embolism
* History of syncope
* Severe anemia
* Abnormal thyroid function
* Severe pulmonary diseases
* Mental illnesses
* Osteoarticular or muscular diseases that impede rehabilitation training

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in VO₂ peak (a marker of cardiopulmonary exercise tolerance) between the two groups before and after 6 months of treatment | At baseline and 6 months after treatment initiation.
  Compare the change in peak oxygen uptake (VO₂ peak, unit: mL/kg/min) between the Exercise Rehabilitation Group and the Basic Treatment Group. VO₂ peak will be measured via cardiopulmonary exercise test at baseline (before treatment initiation) and 6 months after treatment initiation to assess changes in cardiopulmonary exercise tolerance.
Difference in 6-minute walk test (6MWT) distance (a marker of cardiopulmonary exercise tolerance) between the two groups before and after 6 months of treatment | At baseline and 6 months after treatment initiation.
  Compare the change in 6MWT distance (unit: meters) between the Exercise Rehabilitation Group and the Basic Treatment Group. 6MWT will be conducted according to standard clinical protocols at baseline (before treatment initiation) and 6 months after treatment initiation to evaluate changes in functional exercise capacity (a key component of cardiopulmonary exercise tolerance).
Differences in estimated Glomerular Filtration Rate (eGFR) between the two groups before and after 6 months of treatment | At baseline and 6 months after treatment initiation.
  Compare the changes in eGFR (a key indicator of overall renal filtration function) between the Exercise Rehabilitation Group and Basic Treatment Group, to assess the intervention's effect on renal filtration function. Higher eGFR values indicate better renal filtration function.
  Measurement Details: eGFR (unit: mL/min/1.73m²), calculated via the CKD-EPI equation using serum creatinine values measured by standard clinical laboratory biochemical analysis (e.g., enzymatic method).
Difference in Serum Creatinine (Scr) between the two groups before and after 6 months of treatment | At baseline and 6 months after treatment initiation.
  Compare the changes in Scr (a marker of renal excretory function) between the Exercise Rehabilitation Group and Basic Treatment Group, to assess the intervention's effect on renal excretory function. Higher Scr values typically indicate impaired renal excretory function.
  Measurement Details: Scr (unit: μmol/L), measured via standard clinical laboratory biochemical analysis (e.g., picric acid method or enzymatic method).
Difference in Left Ventricular Ejection Fraction (LVEF) between the two groups before and after 6 months of treatment | At baseline and 6 months after treatment initiation.
  Compare the change in Left Ventricular Ejection Fraction (LVEF) between the Exercise Rehabilitation Group and the Basic Treatment Group.Measurement name: Left Ventricular Ejection Fraction (LVEF).Measurement tool: Transthoracic Echocardiography (TTE, standard clinical ultrasound examination).Unit of measure: Percentage (%).Outcome interpretation: Higher LVEF values indicate better left ventricular systolic function (normal range: 50%-70% in adults); changes in LVEF reflect the intervention's effect on cardiac contractile function.LVEF will be measured via TTE at baseline (before treatment initiation) and 6 months after treatment initiation.

SECONDARY OUTCOMES:
Difference in N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels between the two groups before and after 6 months of treatment | At baseline and 6 months after treatment initiation.
  Compare the change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels between the Exercise Rehabilitation Group and the Basic Treatment Group.
  Measurement name: N-terminal pro-B-type natriuretic peptide (NT-proBNP) Measurement tool: Standard laboratory immunoassay (e.g., chemiluminescent immunoassay) Unit of measure: Picograms per milliliter (pg/mL) Outcome interpretation: NT-proBNP is a marker of cardiac wall stress and heart failure severity; lower levels indicate improved cardiac load and reduced heart failure burden.
  Levels will be measured via venous blood sampling at baseline (before treatment initiation) and 6 months after treatment initiation.
Difference in cystatin C (Cys-C) levels between the two groups before and after 6 months of treatment | At baseline and 6 months after treatment initiation.
  Compare the change in cystatin C (Cys-C) levels between the Exercise Rehabilitation Group and the Basic Treatment Group.
  Measurement name: Cystatin C (Cys-C) Measurement tool: Standard laboratory immunoassay (e.g., particle-enhanced turbidimetric immunoassay) Unit of measure: Milligrams per liter (mg/L) Outcome interpretation: Cys-C is a sensitive marker of early renal function impairment; lower levels indicate better glomerular filtration function.
  Levels will be measured via venous blood sampling at baseline (before treatment initiation) and 6 months after treatment initiation.
Difference in high-sensitivity C-reactive protein (hs-CRP) levels between the two groups before and after 6 months of treatment | At baseline and 6 months after treatment initiation.
  Compare the change in high-sensitivity C-reactive protein (hs-CRP) levels between the Exercise Rehabilitation Group and the Basic Treatment Group.
  Measurement name: High-sensitivity C-reactive protein (hs-CRP) Measurement tool: Standard laboratory immunoassay (e.g., latex-enhanced immunoturbidimetry) Unit of measure: Milligrams per liter (mg/L) Outcome interpretation: hs-CRP is a marker of systemic inflammation (closely associated with CRS progression); lower levels indicate reduced inflammatory burden and potential slowing of cardiorenal damage.
  Levels will be measured via venous blood sampling at baseline (before treatment initiation) and 6 months after treatment initiation.
Differences in scores of the Minnesota Living with Heart Failure Questionnaire between the two groups before and after 6 months of treatment | At baseline and 6 months after treatment initiation.
  Compare the change in scores of the Minnesota Living with Heart Failure Questionnaire (MLHFQ) between the Exercise Rehabilitation Group and the Basic Treatment Group, to evaluate the intervention's impact on patients' heart failure-related quality of life.
  Unabbreviated scale title: Minnesota Living with Heart Failure Questionnaire Score range: Minimum value = 0 points, Maximum value = 105 points Outcome interpretation: Higher scores indicate worse quality of life (reflecting more severe heart failure symptoms, greater functional limitations, and increased emotional distress related to the disease); lower scores indicate better quality of life.
  The questionnaire will be completed by participants independently (with researcher assistance if needed for clarity) at baseline (before treatment initiation) and 6 months after treatment initiation, following standard administration guidelines.